CLINICAL TRIAL: NCT05346991
Title: Disseminating an Evidence-based Tobacco Control Intervention for School Teachers in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glorian Sorensen (Other)
Collaborators: Healis-Sekhsaria Institute for Public Health (Other)
Responsible Party: Sponsor-Investigator, Glorian Sorensen, Professor of Social and Behavioral Sciences, Harvard School of Public Health (HSPH)
Organization: Harvard School of Public Health (HSPH) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB16-1055
Record Dates: First submitted 2022-04-15; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Implementation of the Tobacco-Free Teachers, Tobacco Free Society program in government schools in Bihar, India
  Interventions: Other: Tobacco Free Teachers, Tobacco Free Society program
- Control arm (No Intervention): Delayed intervention - control arm schools receive the program after all data collection is complete

INTERVENTIONS:
Other: Tobacco Free Teachers, Tobacco Free Society program — The Tobacco Free Teachers, Tobacco Free Society (TFT-TFS) program provides teachers with the knowledge and skills to quit tobacco use, or to help someone else quit; it also helps schools comply with national tobacco control policies. School principals implement four TFT-TFS program components with teachers in their schools during school hours across an academic year (August-April):
  * Adopting a school tobacco control policy
  * Providing cessation support (e.g. distribution of self-help quit booklets and referrals to government cessation resources)
  * Conducting monthly group discussions with teachers about tobacco
  * Hanging six thematic posters in the school
  With the goal of establishing a tobacco-free school environment, the program incorporates six program themes: 1. Teachers as Role Models; 2. Health Effects of Tobacco; 3. Motivation to Quit-or Help Others to Quit; 4. Skills to Quit; 5. Dealing with Withdrawal; and 6. Maintenance and Celebration.
  Arms: Intervention arm

SUMMARY:
Disseminating an evidence-based tobacco control intervention for School Teachers

DETAILED DESCRIPTION:
There is a profound need for evidence-based interventions that promote tobacco control on a large scale, particularly in low- and middle-income countries. In India in 2010 alone, tobacco use accounted for over one million deaths. The overall goal of this study is to identify effective strategies for broad-based implementation of evidence-based tobacco control interventions that can be embedded in existing organizational infrastructures and accommodate the realities of low-resource settings. This study builds on an intervention for school teachers, called the Tobacco-Free Teachers/Tobacco-Free Society (TFT-TFS) program, shown to be efficacious in increasing tobacco use cessation and tobacco policy implementation in a cluster randomized controlled trial in the Bihar School Teachers' Study (BSTS). Teachers in India are an important channel for promoting tobacco control, given their roles as community leaders and role models. The next logical step in this research is to develop the knowledge, products and processes needed to take this intervention to scale and disseminate it through readily accessible and sustainable channels. Investigators will test an implementation model for building capacity within education departments to support and deliver this program within schools, using the existing infrastructure for curriculum training in state education departments. Within each state in India, schools are organized within clusters, and cluster coordinators are responsible for directly training principals about curriculum issues. The investigators will build the capacity of cluster coordinators to train and support principals in implementing the TFT-TFS program in their schools. The central research question of this study is: Will this evidence-based intervention be successfully adopted, implemented, and sustained through existing channels using this implementation process? The specific aims are to: (1) determine the extent to which this implementation model meets acceptable rates of program adoption, implementation, reach and maintenance of the TFT-TFS program among schools in the Indian state of Bihar; (2) determine program effectiveness in increasing tobacco use cessation and implementation of tobacco control policies in schools; (3) determine the feasibility of building the capacity of cluster coordinators to train and support principals in program implementation and maintenance in schools, and for the Department of Education to sustain the program; and (4) determine the direct financial costs of program implementation and maintenance. This study uses a non-inferiority design to test the primary hypothesis that program adoption, implementation, and reach will not be inferior to the high standards demonstrated in BSTS; and assesses program effectiveness in improving tobacco use cessation and increasing policy implementation using a cluster randomized design. This research is innovative because it systematically examines the process of scaling up one of the first evidence-based approaches to tobacco use cessation among adults in India. This study is significant because it is expected to improve understanding of implementation processes needed for taking evidence-based interventions to scale.

ELIGIBILITY:
Inclusion Criteria:

* All teachers and principals employed in intervention and control schools

Exclusion Criteria:

* None

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1102 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Tobacco use cessation among teachers | Immediately post-intervention
  Self-administered Teacher's Survey completed by teachers. Using survey data, compute 7- and 30-day quit prevalence among teachers who reported using any tobacco in the last 9 months (the length of the academic year), and compare measures between intervention and control schools

SECONDARY OUTCOMES:
School tobacco control policy implementation - School Observation | Immediately post-intervention
  School Observation Checklist completed by an independent evaluator. Observations include the number of physical locations in the school and grounds with evidence of tobacco use (range 0 - 10, lower score indicates less evidence of tobacco use).
School tobacco control policy implementation - Teachers' Report | Immediately post-intervention
  Self-administered Teacher's Survey completed by teachers. Using survey data, compute a composite score of five questions regarding presence of a tobacco policy and it's enforcement at the school (range 0-5, higher score indicates stricter policy.

CONTACTS AND LOCATIONS:
Overall Officials: Glorian Sorensen, PhD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States
- Healis Sekhsaria Institute for Public Health, Mumbai, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nagler EM, Pednekar M, Sinha DN, Stoddard AM, Narake S, Adhikari K, Jones L, Lando H, Vriniotis M, Gupta P, Sorensen G. Implementation of an evidence-based tobacco control intervention for school teachers in India: Evaluating the effects of a capacity-building strategy. Implement Res Pract. 2023 Mar 22;4:26334895231159428. doi: 10.1177/26334895231159428. eCollection 2023 Jan-Dec. PMID 37091538